CLINICAL TRIAL: NCT00981045
Title: Randomized Evaluation of Efficacy and Safety of Ferric Carboxymaltose in Patients With Iron Deficiency Anemia and Impaired Renal Function
Brief Title: Evaluation of Efficacy and Safety of Ferric Carboxymaltose (FCM) in Patients With Iron Deficiency Anemia and Impaired Renal Function
Acronym: REPAIR-IDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT09030
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency Anemia; Impaired Renal Function
Keywords: IDA
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): 2 doses at 15 mg/kg to a maximum 750 mg per dose for a total maximum cumulative dose of 1500 mg
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Iron Sucrose (Venofer) (Active Comparator): 5 doses of 200 mg for a total cumulative dose of 1000 mg
  Interventions: Drug: Iron Sucrose (Venofer)

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — 2 doses at 15 mg/kg to a maximum 750 mg per dose for a total maximum cumulative dose of 1500 mg
  Arms: Ferric Carboxymaltose (FCM)
Drug: Iron Sucrose (Venofer) — 5 doses of 200 mg for a total cumulative dose of 1000 mg
  Arms: Iron Sucrose (Venofer)

SUMMARY:
The primary objective of this study is to examine the efficacy and safety (cardiovascular) of an investigational intravenous (IV) iron, ferric carboxymaltose (FCM), compared to IV iron sucrose (Venofer) in subjects who have iron deficiency anemia (IDA) and impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > or = to 18 years of age.
* Chronically impaired renal function.
* Screening visit central laboratory hemoglobin < or = to 11.5 g/dL.
* Screening ferritin < or = to 100 ng/mL or < or = to 300 when transferrin saturation (TSAT) is < or = to 30%.
* If on an erythropoiesis stimulating agent(ESA) a stable dose (+/- 20%) for 4 weeks prior to randomization.

Exclusion Criteria:

* Known hypersensitivity reaction to any component of ferric carboxymaltose (FCM) or Venofer.
* Previously randomized in a clinical study of Ferric Carboxymaltose (FCM).
* Requires dialysis for treatment of chronic kidney disease OR is being considered for initiation of dialysis during the time period of this trial.
* No evidence of iron deficiency.
* Any non-viral infection.
* AST or ALT at screening as determined by central labs greater than 1.5 times the upper limit of normal.
* Known positive hepatitis with evidence of active disease.
* Received an investigational drug within 30 days of screening.
* Alcohol or drug abuse within the past 6 months.
* Hemochromatosis or other iron storage disorders.
* Estimated life expectancy of less than 6 months, or for cancer patients, an ECOG Performance Status greater than 1.
* Any other laboratory abnormality, medical condition or psychiatric disorder which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements.
* Pregnant or sexually-active female subjects who are not willing to use an acceptable form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2561 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 04-Sept-2009 through 15-Jun-2011; Hospitals and Medical Clinics
Pre-assignment Details: 14 subjects randomized to FCM and 9 subjects randomized to Venofer were discontinued prior to dosing due to subject request or selection criteria/study compliance reasons.
Groups:
- Ferric Carboxymaltose (FCM): Ferric Carboxymaltose (FCM) : 2 doses at 15 mg/kg to a maximum 750 mg per dose for a total maximum cumulative dose of 1500 mg
- Iron Sucrose (Venofer): Iron Sucrose (Venofer) : 5 doses of 200 mg for a total cumulative dose of 1000 mg
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (Venofer)
Started | 1290 | 1294
Completed | 1276 | 1285
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Population: 14 subjects randomized to receive FCM and 9 subjects randomized to receive Venefor were randomized but discontinued prior to dosing due to subject request or selection criteria/study compliance reasons.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (Venofer) | Total
Number analyzed (Participants) | 1276 | 1285 | 2561
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 468 | 500 | 968
  >=65 years | 808 | 785 | 1593
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (13.00) | 67.2 (13.00) | 67.3 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 810 | 818 | 1628
  Male | 466 | 467 | 933
Region of Enrollment [Number; unit: participants]
  United States | 1276 | 1285 | 2561

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the Highest Observed Hemoglobin Any Time From Baseline to End of Study.
Time Frame: Day 56
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (Venofer)
Number analyzed (Participants) | 1249 | 1244
g/dL | 1.13 (1.044) | 0.92 (0.917)

2. Primary Outcome: Proportion of Subjects Experiencing at Least One Event in the Primary Composite Safety Endpoint in the Randomized Population.
Description: The primary composite safety endpoint was defined as death due to any cause, nonfatal myocardial infarction, nonfatal stroke, unstable angina requiring hospitalization or medical intervention, arrhythmias, protocol-defined hypersensitive events, and protocol-defined hyposensitive events.
Time Frame: Day 120
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (Venofer)
Number analyzed (Participants) | 1276 | 1285
participants | 175 | 156

ADVERSE EVENTS:
Time Frame: September 4, 2009 through June 15, 2011
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (Venofer)
Serious Adverse Events (participants affected / at risk) | 202/1276 | 197/1285
Other Adverse Events (participants affected / at risk) | 305/1276 | 151/1285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=1276) | Iron Sucrose (Venofer) (N=1285)
Anemia (Blood and lymphatic system disorders) | 14 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 6 | 11
Angina pectoris (Cardiac disorders) | 6 | 3
Angina unstable (Cardiac disorders) | 6 | 3
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 2
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bifascicular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 4
Cardiac arrest (Cardiac disorders) | 0 | 4
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 30 | 29
Cardio-respiratory arrest (Cardiac disorders) | 2 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 5 | 3
Ischemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 5
Myocardial ischemia (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Superventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Retinal vein occlusion (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Fecaloma (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis hemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 9 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal ischemia (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intra-abdominal hematoma (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 3
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 4
Fatigue (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 1
Generalized edema (General disorders) | 1 | 2
Hernia obstructive (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 3
Edema peripheral (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Ulcer hemorrhage (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Pancreas transplant rejection (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bacteremia (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 10 | 6
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 5 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 1
Osteomyelitis (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 15 | 16
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Renal cyst infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal bacteremia (Infections and infestations) | 0 | 1
Staphy;ococcal infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 10 | 2
Urosepsis (Infections and infestations) | 0 | 3
Wound infection (Infections and infestations) | 1 | 0
Device lead damage (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1
Liver function abnormal (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 6
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycemic coma (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 5
Syncope vasovagal (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 4
Delirium (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status change (Psychiatric disorders) | 2 | 1
Azotemia (Renal and urinary disorders) | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 2 | 0
Renal artery occlusion (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 8
Renal failure acute (Renal and urinary disorders) | 13 | 11
Renal failure chronic (Renal and urinary disorders) | 10 | 10
Renal impairment (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Angiedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 2
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=1276) | Iron Sucrose (Venofer) (N=1285)
Hypertension (Vascular disorders) | 133 | 95
Nausea (Gastrointestinal disorders) | 172 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less